CLINICAL TRIAL: NCT06505369
Title: A Phase II Study Measuring MRD Negativity After Bispecific T-cell Redirectors Talquetamab and Teclistamab Consolidation in Sequence as Part of First Line Treatment in Transplant Eligible Multiple Myeloma Patients
Brief Title: Bispecific T-cell Redirectors as Part of First Line Treatment in Transplant Eligible Multiple Myeloma Patients
Acronym: TALTEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: North Estonia Medical Centre (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CT number 2023-508212-38-00
Record Dates: First submitted 2024-06-18; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Transplant Eligible; Talquetamab; Teclistamab; MRD negativity
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone; talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction with Dara -VRd + Consolidation with Talquetamab and Teclistamab as monotherapy in sequence (Experimental): Induction with Daratumumab-VRd; Consolidation part I with Talquetamab; Consolidation part II with Teclistamab.
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Talquetamab; Drug: Teclistamab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered by SC injection
  Other Names: JNJ-54767414
Drug: Bortezomib — Bortezomib will be administered by SC injection
  Other Names: EU Substance number SUB20020
Drug: Lenalidomide — Lenalidomide will be administered by oral route
  Other Names: EU Substance number SUB25389
Drug: Dexamethasone — Dexamethasone will be administered by oral route
  Other Names: EU Substance number SUB07017MIG
Drug: Talquetamab — Talquetamab will be administered by SC injection
  Other Names: JNJ-64407564
Drug: Teclistamab — Teclistamab will be administered by SC injection
  Other Names: JNJ-64007957

SUMMARY:
This is Phase 2, open-label, multicentre, non-randomised study evaluating participants with newly diagnosed MM eligible for high-dose therapy. The goal of the study is to determine if consolidation with T-cell redirectors - Talquetamab and Teclistamab in sequence will improve the response depth: increase MRD negative CR rate.

DETAILED DESCRIPTION:
A total of 50 transplant-eligible patients with newly diagnosed multiple myeloma in need of treatment will be enrolled.

The study consists of three phases: Induction, Consolidation, and Follow-up. Induction will consist of Dara-VRd and consolidation Part I will include talquetamab and Part II will include teclistamab.

Follow-up Phase After consolidation, treatment continues upon physician's choice: the options are ASCT with maintenance or only maintenance with lenalidomide.

Efficacy will be evaluated by serum/urine electrophoresis monthly; by serum/urine immunofixation, bone marrow morphology and flow cytometry when CR/sCR is suspected;

MRD will be evaluated by NGS ( at the level of 10-6) and FDG PET-CT ( by Deauville score) at various timepoints during induction, consolidation and follow-up.

Participants quality of life, symptoms, functional and general well-being will be captured using 3 PRO measures ( PRO-CTCAE, EORTC QLQ-C30, FACT-Cog).

The safety of study drugs will be assessed by physical examinations, vital signs, ECGs, clinical laboratory tests, neurologic examinations (including ICE scores), ECOG performance status, and AE monitoring according to NCI-CTCAE Version 5.0), grading of CRS and ICANS will be assessed based on ASTCT guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have documented MM satisfying the IMWG criteria.
2. Newly diagnosed patients eligible for high dose therapy and ASCT.
3. ECOG performance status score ≤2.
4. HIV-positive participants are eligible if they meet all of the following

   1. No detectable viral load (ie, <50 copies/mL) at screening
   2. CD4+ count >300 cells/mm3 at screening
   3. No AIDS-defining opportunistic infection within 6 months of screening
   4. Receiving HAART. Any changes in HAART due to resistance/progression should occur at least 3 months prior to screening. A change in HAART due to toxicity is allowed up to 4 weeks prior to screening.
5. Must sign an ICF indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.
6. Willing and able to adhere to the lifestyle restrictions specified in this protocol.
7. A female participant of childbearing potential must have a negative highly sensitive serum (β hCG) pregnancy test at screening
8. A female participant must be

   1. Not of childbearing potential or
   2. Of childbearing potential and practicing true abstinence; or have a sole partner who is vasectomized; or practicing 2 effective methods of contraception
9. A female participant must agree not to donate eggs or freeze for future use during the study and for 6 months after receiving the last dose of study treatment.
10. A male participant must wear a condom when engaging any sexual activity that allows for passage of ejaculate to another person during the study and for a minimum of 100 days after receiving the last dose of study treatment.
11. A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 100 days after receiving the last dose of study treatment.
12. Have clinical laboratory values meeting the following criteria

    1. Hemoglobin ≥8 g/dL
    2. Platelets ≥75×109/L
    3. ANC ≥1.0×109/L
    4. AST and ALT ≤2.5×ULN
    5. eGFR ≥30 mL/min
    6. Total bilirubin <1.5×ULN

Exclusion Criteria:

1. Waldenström's macroglobulinemia, POEMS syndrome, or primary amyloid light chain amyloidosis.
2. Known active CNS involvement or exhibits clinical signs of meningeal involvement of MM. If either is suspected, negative whole brain MRI and lumbar cytology are required.
3. Peripheral neuropathy or neuropathic pain Grade 2 or higher
4. Excluded for any of the following:

   1. Any ongoing myelodysplastic syndrome or B cell malignancy (other than MM).
   2. Any history of malignancy, other than MM, which is considered at high risk of recurrence requiring systemic therapy.
   3. Any active malignancy (ie, progressing or requiring treatment change in the last 24 months) other than MM. The only allowed exceptions are malignancies treated within the last 24 months that are considered cured:

      1. Non-muscle invasive bladder cancer (solitary Ta-PUN-LMP or low grade, <3 cm, no CIS).
      2. Non-melanoma skin cancers treated with curative therapy or localized melanoma treated with curative surgical resection alone.
      3. Non-invasive cervical cancer.
      4. Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ or history of localized breast cancer (anti-hormonal therapy is permitted).
      5. Localized prostate cancer (M0, N0) with a Gleason Score ≤7a, treated locally only (RP/RT/focal treatment).
      6. Other malignancy that is considered cured with minimal risk of recurrence in consultation with the sponsor's medical monitor.
5. Stroke within 6 months prior to signing ICF.
6. Presence of the following cardiac conditions:

   1. New York Heart Association stage III or IV congestive heart failure (see Appendix )
   2. Myocardial infarction or coronary artery bypass graft ≤6 months prior to enrollment, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina)
   3. Uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities
   4. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
   5. History of severe non-ischemic cardiomyopathy
7. Concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study, such as:

   1. Uncontrolled diabetes
   2. Evidence of active systemic viral, fungal, or bacterial infection, requiring systemic antimicrobial therapy
   3. History of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing
   4. Gastrointestinal disease that may significantly alter the absorption of oral drugs
   5. Disabling psychiatric conditions (eg, alcohol or drug abuse), severe dementia, or altered mental status
8. Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
9. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients
10. Any of the following:

    1. Hepatitis B infection (ie, HBsAg or HBV-DNA positive).
    2. Active hepatitis C infection as measured by positive HCV-RNA testing.
11. Prior or current systemic therapy or stem cell transplantation for any plasma cell dyscrasia, with the exception of emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
12. Major surgery within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment.
13. Contraindications to the use of Dara-VRd per SmPC.
14. Prior or concurrent exposure to any of the following, in the specified time frame prior to first dose of study treatment:

    1. Investigational vaccine other than SARS-CoV-2 vaccine approved/in use under emergency approval within 4 weeks. Non-live or non-replicating vaccines authorized for emergency use (eg, COVID-19) by local health authorities are allowed.
    2. Live, attenuated vaccine within 4 weeks
    3. Monoclonal antibody therapy within 21 days (not used for the treatment of MM)
    4. Received a strong CYP3A4 inducer within 5 half-lives prior to start of administration of study treatment
15. Participant is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of study treatment.
16. Participant plans to father a child while enrolled in this study or within 100 days after the last dose of study treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission rate by next generation sequencing ( NGS) after completing consolidation with talquetamab and teclistamab. | 18 months approximately
  MRD measured by NGS with a sensitivity level of 10-6.
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission rate by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan after completing consolidation with talquetamab and teclistamab. | 18 months approximately
  MRD assessed by FDG PET-CT scan using Deauville score.

SECONDARY OUTCOMES:
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission rate by next generation sequencing ( NGS) after completing induction treatment with Daratumumab-VRd | 6 months approximately
  MRD measured by NGS with a sensitivity level of 10-6.
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission rate by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan after completing induction treatment with Daratumumab-VRd. | 6 months approximately
  MRD assessed by FDG PET-CT scan using Deauville score.
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission conversion by next generation sequencing ( NGS) after completing consolidation treatment with talquetamab. | 12 months approximately
  MRD measured by NGS with a sensitivity level of 10-6.
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission conversion by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan after completing consolidation treatment with talquetamab. | 12 months approximately
  MRD assessed by FDG PET-CT scan using Deauville score.
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission conversion by next generation sequencing ( NGS) after completing consolidation treatment with teclistamab. | 18 months approximately
  MRD measured by NGS with a sensitivity level of 10-6.
Evaluate efficacy in terms of Minimal Residual Disease (MRD) negative Complete Remission conversion by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan after completing consolidation treatment with teclistamab. | 18 months approximately
  MRD assessed by FDG PET-CT scan using Deauville score.
Evaluate efficacy in terms of Sustained Minimal Residual Disease (MRD) negative Complete Remission rate by next generation sequencing ( NGS). | 42 months approximately
  MRD measured by NGS with a sensitivity level of 10-6.
Evaluate efficacy in terms of Sustained Minimal Residual Disease (MRD) negative Complete Remission rate by Fluorodeoxyglucose Positron Emission Tomography-Computerized Tomography (FDG PET-CT) scan. | 42 months approximately
  MRD assessed by FDG PET-CT scan using Deauville score.
To assess Overall Response Rate (ORR) | 42 months approximately
  ORR is defined as proportion of patients achieveing documentation of a response (Partial Response or better) from the first dose of study drug on treatment. Response to treatment is defined according to the International Myeloma Working Group (IMWG) criteria.
To assess Overall Survival (OS). | 42 months approximately
  OS is defined as the time from the date of first dose of study drug to the date of the subject's death. If the subject is alive or the vital status is unknown, then the subject's data will be censored at the date the subject was last known to be alive. OS is measured in months.
To assess Progression free Survival (PFS). | 42 months approximately
  PFS is defined as the time from the date of first dose of study drug to the date of first documented disease progression, as defined in the International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first. For subjects who have not progressed and are alive, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy. PFS is measured in months.
To assess Duration of Response ( DoR). | 42 months approximately
  DoR is the date of initial documentation of a response (Partial Response or better) to the date of first documented evidence of progressive disease, as defined in the International Myeloma Working Group (IMWG) criteria. Relapse from complete response is not considered as disease progression. For subjects who have not progressed, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy. DoR is measured in months.
To assess Time to Next anti-myeloma Treatment (TNT). | 42 months approximately
  TNT is defined as the time between date of first dose of study drug and the first dose of the next treatment received. TNT is measured in months.
To assess the safety and tolerability of the treatment described in the protocol. | 42 months approximately
  Incidence of treatment-emergent adverse events. AE monitoring according to NCI-CTCAE Version 5.0), grading of CRS and ICANS will be assessed based on ASTCT guidelines.
To assess quality of life on the treatment described in the protocol. | 42 months approximately
  Quality of life in general is assessed using PRO questionnaire, such as EORTC QLQ-C30.
To assess incidence of participant -recorded side effects on the treatment described in the protocol. | 42 months approximately
  Participant - recorded side effects are assessed using PRO questionnaire, such as PRO-CTCAE.

OTHER OUTCOMES:
To capture specific proteomic signatures from MRD positive and negative patients by mass-spectrometry based proteomic profiling. | 42 months approximately

CONTACTS AND LOCATIONS:
Overall Officials: Diana Loigom, MD, Principal Investigator — North Estonia Medical Centre
Locations (7):
- Denmark (3):
  - Copenhagen University Hospital (Rigshospitalet), Copenhagen
  - Odense University Hospital, Odense
  - Vejle hospital, Vejle
- North Estonia Medical Centre, Tallinn, Estonia
- Norway (3):
  - Oslo University Hospital, Oslo Myeloma Centre, Oslo
  - Stavanger University Hospital, Stavanger
  - St. Olavs Hospital, Trondheim